CLINICAL TRIAL: NCT02812524
Title: Intratumoral Ipilimumab in Head and Neck Cancer
Brief Title: Ipilimumab for Head and Neck Cancer Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-042
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Immunotherapy; Yervoy; Head and neck cancer; Pre-operative
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intratumoral Ipilimumab (Experimental): Patients receive a 3mg intratumoral injection of ipilimumab during a biopsy procedure.
  Interventions: Drug: Intratumoral Ipilimumab

INTERVENTIONS:
Drug: Intratumoral Ipilimumab — Patients with a planned resection of SCCHN will have a biopsy procedure 7-10 days prior to surgery and receive an injection of ipilimumab directly into a tumor.
  Other Names: Yervoy; BMS734016; MDX-010

SUMMARY:
This study is for patients with squamous cell carcinoma of the head and neck (SCCHN). This study will test the feasibility of the administration of intratumoral injections of ipilimumab prior to surgical resection, and the immune system response to treatment.

DETAILED DESCRIPTION:
This study will test intratumor microdosing of ipilimumab (antagonistic antibody directed to Cytotoxic T-Lmphocyte-Associated Protein 4 [CTLA-4]) 7-10 days prior to planned surgical resection of tumor and involved lymph nodes in patients with SCCHN. Tissue, peripheral blood, saliva and stool samples will be obtained for immunologic end points. The primary objective is to assess safety, as determined by the number of surgeries that are delayed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SCCHN who are planned for surgical resection and in the opinion of the surgeon are able to safely undergo tissue biopsy plus intratumoral (IT) injection in advance, with special consideration given to risk of occlusion or compression of airway or major vessels in the neck, secondary to tumor swelling, or erosion into a major vessel in the case of necrosis.
* Age 18 years or above with ability to give informed consent, comply with the protocol and sign a study-specific consent document. Patients with history of psychiatric illness must be judged by the investigator as able to understand the investigational nature and risks associated with the therapy.
* Any Eastern Cooperative Oncology Group (ECOG) performance status deemed suitable by investigator for requirements of study, to potentially include incisional office biopsy of lesion, or image guided multiple 18g core needle biopsies (5 minimum) by interventional radiology, followed immediately by direct injection of lesion with drug.
* Patients must have blood test results within protocol-specified parameters
* Men must agree to not attempt to become a new father for a total of 165 days post-treatment completion
* Women must agree not to become pregnant for a total of 105 days post treatment completion

Exclusion Criteria:

* Any clinical factors such as bleeding, active infection, colitis history or psychiatric factors that in the judgment of the investigator would preclude safe participation and compliance with study procedures.
* Need for chronic maintenance oral steroids ≥ 20mg prednisone daily equivalent; inhaled steroids are acceptable.
* History of or current active autoimmune diseases, [e.g. including but not limited to inflammatory bowel diseases (IBD), rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barre syndrome), which in the judgment of the investigator pose an active and significant risk. Vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are not exclusionary.]
* Infectious diseases including human immunodeficiency virus (HIV), Hepatitis B virus (HBV) and hepatitis C virus (HCV).
* Patients who have had a history of acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation, and in the judgment of the investigator still pose an active risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Surgery delay | 7-10 Days
  The percentage of patients with surgery delayed possibly related to the study drug.

SECONDARY OUTCOMES:
Feasibility of paired tissue sample acquisition | 7-10 Days
  The number of tissue samples that can be collected which were: biopsied, injected, and resected.
Acceptance of study | 28 Days
  The screening-to-enrollment ratio will be calculated.

OTHER OUTCOMES:
Failure rate of planned laboratory assays | 7-10 days
  The percentage of assays achieving a result.

CONTACTS AND LOCATIONS:
Overall Officials: Rom S Leidner, MD, Principal Investigator — Providence Health & Services; R. Bryan Bell, MD, DDS, Principal Investigator — Providence Health & Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — https://oregon.providence.org/our-services/p/providence-cancer-center/